CLINICAL TRIAL: NCT00157287
Title: A Cluster Randomized Trial to Improve Weaning and Extubation From Mechanical Ventilation in Community Hospitals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-01-076
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Evidence based weaning protocol

SUMMARY:
Protocol directed weaning has been shown to reduce the duration of mechanical ventilation for patients admitted to the intensive care unit (ICU) of tertiary centres. However, this benefit has not previously been studied in a community hospital setting. We therefore sought to evaluate the impact of an evidence-based weaning guideline on the outcomes for patients receiving mechanical ventilation in the ICUs of community hospitals in a cluster randomized controlled trial involving 11 community hospitals.

ELIGIBILITY:
Inclusion Criteria:

* patients ventilated for more than 24 hours

Exclusion Criteria:

* patients less than 16 years of age patients who receive only non-invasive ventilation patients chronically ventilated at time of ICU admission patients who will not be candidates for weaning from ventilation at time of admission If withdrawl of life support is imminent at the point the patient has been ventilated for 24 hours

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2005-06 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
ICU length of stay

SECONDARY OUTCOMES:
duration of ventilation
length of hospital stay
complications (re-intubation within 48 hours, pneumonia within 48 hours)
ICU mortality
Hospital mortality
ICU readmissions
Qulaity of life

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Butler, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Claudio Martin, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Femida Gwadry-Sridhar, MSc, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (11):
- Canada (11):
  - William Osler Health Centre (Brampton), Brampton, Ontario
  - Brant Community Health Systems, Brantford, Ontario
  - Joseph Brant Memorial Hospital, Burlington, Ontario
  - Guelph General Hospital, Guelph, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - North Bay General Hospital, North Bay, Ontario
  - Lakeridge Health Corporation (Oshawa), Oshawa, Ontario
  - Stratford General Hospital, Stratford, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Hotel Dieu of St. Joseph, Windsor, Ontario